CLINICAL TRIAL: NCT02837887
Title: A Computerized Cognitive Behavioral Therapy for Cancer Patients With Major Depressive Disorder
Brief Title: Computerized Cognitive Behavior Therapy in Treating Depression in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Barbara Andersen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-16008; NCI-2016-00954 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Major Depressive Disorder
Keywords: Cancer; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Neoplasms; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (immediate treatment) (Experimental): Patients undergo computerized cognitive behavior therapy consisting of 45-60 minute sessions once per week for 8 weeks. Patients also complete the PHQ-9 and GAD7 at weeks 1, 3, 5, 7 and 8 and complete other questionnaires for 15-30 minutes each that assess psychosocial and physical symptoms.
  Interventions: Behavioral: Computerized Cognitive Behavior Therapy
- Group II (wait-list) (Experimental): Patients are placed on an 8-week wait-list and then undergo computerized cognitive behavior therapy and receive questionnaires as in Group I.
  Interventions: Behavioral: Computerized Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Computerized Cognitive Behavior Therapy — Undergo computerized cognitive behavior therapy
  Other Names: cCBT; cognitive behavior therapy; Beating the Blues; CBT

SUMMARY:
This randomized clinical trial studies how well a computerized cognitive behavior therapy program works in treating depression in patients with cancer. The cognitive behavior therapy program uses a series of internet-delivered sessions intended to help patients identify and change problematic patterns of thinking and behavior that maintain depression.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the efficacy of computerized cognitive behavior therapy ("Beating the Blues") in reducing symptoms of depression and remission of major depressive disorder (MDD) in cancer patients.

II. Test the feasibility of implementation and patient acceptability of online computerized cognitive behavior therapy for cancer patients with major depressive disorder (MDD).

III. Test moderators (cancer specific stress, MDD history, anxiety disorder comorbidity, and homework compliance) of treatment outcome.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (IMMEDIATE TREATMENT): Patients undergo computerized cognitive behavior therapy consisting of 45-60 minute sessions once per week for 8 weeks. Patients also complete the Patient Health Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder-7 (GAD7) at weeks 1, 3, 5, 7 and 8 and complete other questionnaires for 15-30 minutes each that assess psychosocial and physical symptoms.

GROUP II (WAIT-LIST): Patients are placed on an 8-week wait-list and then undergo computerized behavior therapy and receive questionnaires as in Group I.

After completion of study intervention, patients are followed up at 2, 4, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* A current/prior cancer diagnosis
* A principal diagnosis of major depressive disorder (MDD)
* Able and willing to give informed consent
* Have access to a computer with an internet connection at home

Exclusion Criteria:

* History of bipolar affective disorder or psychosis
* History of substance dependence in the past six months
* Subnormal intellectual potential (intelligence quotient [IQ] below 80)
* Current suicide risk or significant intentional self-harm in the last six months sufficient to preclude treatment on an outpatient basis
* Inability to read and write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Rating Scale for Depression (HRSD) | Week 0 to Week 8
  The 17-item HRSD, modified to assess atypical symptoms, is a standard interview-administered measure of depressive symptom severity. The HRSD will be administered by study personnel supervised by the Principal Investigator.

SECONDARY OUTCOMES:
Change in the Beck Depression Inventory (BDI-II) | Week 0 to week 8
  The PHQ9 is a 9-item self-report measure based on the diagnostic criteria for major depression from the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change in Patient Health Questionnaire-9 (PHQ-9) | Week 0 to week 8
  21 item self report measures of depressive symptoms
Change in Generalized Anxiety Disorder-7 (GAD7) | Week 0 to week 8
  The GAD7 is a 7-item self-report measure based on the diagnostic criteria for generalized anxiety disorder from the DSM-IV.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Andersen, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University, Columbus, Ohio, United States